CLINICAL TRIAL: NCT01751178
Title: Clinical Study to Evaluate the Efficacy of Chlorhexidine Mouthwashes
Brief Title: An Efficacy Study of Chlorhexidine Mouthwashes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RH01561
Record Dates: First submitted 2012-12-13; First posted 2012-12-17 (Estimated); Results first posted 2014-07-28 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-06

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis | interventions — Ethanol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mouthwash with Alcohol (Active Comparator): rinse with 10ml 0.2% w/v Chlorhexidine Digluconate Mouthwash with alcohol for 1 timed minute twice daily for 6 weeks following brushing with a full brush head of standard toothpaste for 1 timed minute.
  Interventions: Drug: Chlorhexidine Digluconate Mouthwash with Alcohol
- Mouthwash without Alcohol (Active Comparator): rinse with 10ml 0.2% w/v Chlorhexidine Digluconate Mouthwash without alcohol for 1 timed minute twice daily for 6 weeks following brushing with a full brush head of standard toothpaste for 1 timed minute.
  Interventions: Drug: Chlorhexidine Digluconate Mouthwash without Alcohol

INTERVENTIONS:
Drug: Chlorhexidine Digluconate Mouthwash with Alcohol — 0.2% w/v Chlorhexidine Digluconate, alcohol containing - UK Marketed Mouthwash
  Arms: Mouthwash with Alcohol
Drug: Chlorhexidine Digluconate Mouthwash without Alcohol — 0.2% w/v Chlorhexidine Digluconate, without alcohol - UK Marketed Mouthwash
  Arms: Mouthwash without Alcohol

SUMMARY:
The aim of this study is to compare subject gingival health after 6 weeks of twice daily use of a non-alcohol or alcohol containing mouthrinse and brushing compared to brushing only.

ELIGIBILITY:
Inclusion Criteria:

* Good general health with (in the opinion of the investigator) no clinically significant and relevant abnormalities of medical history or oral/ dental examination.

  5. a) Good oral health in the opinion of the investigator (allowing mild to moderate gingivitis to meet entry criteria).

  b) A minimum of 20 permanent gradable teeth at screening. (Gradable teeth are those where restorative materials cover less than 25% of the tooth surface graded).

  c) Mild to moderate gingivitis present at the screening visit in the opinion of the investigator.

  d) Positive response to bleeding on brushing exercise at screening visit. e) A total of 20 bleeding sites or greater at baseline visit.

Exclusion Criteria:

* Known or suspected intolerance or hypersensitivity to Chlorhexidine or other study materials (or closely related compounds) or any of their stated ingredients.
* 5. a) Current or relevant history of any serious, severe or unstable physical or psychiatric illness or any other medical condition (e.g. Diabetes Mellitus) that would make the subject unlikely to fully complete the study or any that increases the risk to the subject or undermines the data validity.

  b) Subjects requiring prophylactic antibiotic treatment prior to dental therapy.

  c) Use of concomitant medication that, in the opinion of the investigator, might interfere with the outcome of the study or increases the risk to the subject (eg: phenytoin, calcium antagonists, cyclosporine, warfarin, antibiotics, immuno-suppressants).

  d) Use of antibiotics within two weeks prior to the screening visit or throughout the study.

  e) Use of any systemic medication which would have an effect on gingival conditions within 14 days of gingival examinations (eg: ibuprofen or aspirin therapy) 6. a) Have current active caries b) More than 3 pockets with 5mm or over. c) Excessive calculus present that interferes with the probing examination for Gingival Index.

  d) Other severe oral/ gingival conditions (e.g. Acute Necrotizing Ulcerative Gingivitis) that may compromise the study or the subjects in the opinion of the investigator or gingivitis examiner.

  e) Medical conditions which may directly influence gingival bleeding. f) Restorations in a poor state of repair. g) Orthodontic appliances anterior cosmetic restorations and veneers. h) Enamel pitting/irregularities. 7. Subjects using chewing tobacco, pan, pan-masala, gutkha or other chewing tobacco products or subjects who have quit using any of those within the past six months prior to screening.

  8. b) An employee of any toothpaste manufacturer or their immediate family.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 324 (Actual)
Dates: Start 2012-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United Kingdom (3):
  - Intertek 4-Front Research - Widnes, Widnes, Cheshire
  - 4Front, Ellesmere Port, Cheshire
  - Intertek - Manchester Science Park, Manchester

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the clinical site.
Pre-assignment Details: A total of 775 subjects were screened and 324 subjects were randomised of whom 319 completed the study. The high screen failure rate was due mainly to subjects not having sufficient permanently gradable teeth.
Groups:
- Reference: Brushing alone with the standard toothpaste for one timed minute twice daily for 6 weeks.
Period: Overall Study
Arm/Group | Mouthwash With Alcohol | Mouthwash Without Alcohol | Reference
Started | 108 | 109 | 107
Completed | 105 | 109 | 105
Not Completed | 3 | 0 | 2
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Other Reason (unknown) | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Reference: Brushing alone with the standard toothpaste for 1 timed minute twice daily for 6 weeks.
- Total: Total of all reporting groups
Arm/Group | Mouthwash With Alcohol | Mouthwash Without Alcohol | Reference | Total
Number analyzed (Participants) | 108 | 109 | 107 | 324
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.8 (10.89) | 36.2 (11.31) | 36.5 (10.48) | 36.8 (10.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 79 | 75 | 239
  Male | 23 | 30 | 32 | 85

OUTCOME MEASURES:

1. Primary Outcome: Gingival Severity Index (GSI) Based on the Gingival Index (GI)
Description: Measure of gingival severity averaged across whole mouth site; each site scored 0, 1, 2, 3 based on GI and,
  1. GSI = 0 if GI is 0 or 1 (no bleeding)
  2. GSI = 1 if GI is 1 or 2 (bleeding)
Time Frame: Change from baseline to 6 weeks
Population: This analysis was conducted on the Intent-to-Treat (ITT) population, defined as those subjects who received study treatment and had at least one post-baseline efficacy measurement.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Mouthwash With Alcohol | Mouthwash Without Alcohol | Reference
Number analyzed (Participants) | 105 | 109 | 105
Units on a scale | 0.152 (0.0085) | 0.143 (0.0072) | 0.212 (0.0121)
Statistical Analysis 1: Comparison: Mouthwash With Alcohol vs Reference; Null hypothesis stated that there was no difference between the two groups; Test type: Superiority or Other; p < 0.0001, ANCOVA — From ANCOVA with factors for treatment group, site, smoking status, number of bleeding sites strata and the baseline GSI as a covariate; Adjusted Mean Difference = -0.061, 95% CI 2-sided [-0.081 to -0.041] — Difference is first named treatment minus second named treatment such that a negative difference favours the first named treatment
Statistical Analysis 2: Comparison: Mouthwash Without Alcohol vs Reference; Null hypothesis stated that there was no difference between the two treatment groups; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Adjusted Mean Difference = -0.070, 95% CI 2-sided [-0.090 to -0.050] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Gingival Index
Description: The GI was assessed on the facial and lingual surfaces at six sites on each tooth (facial and lingual - distal papillae, margin and mesial papillae). These assessments were performed on all evaluable teeth using moderate pressure sweeping a blunt ended probe, which was engaged in approximately 1 millimetre (mm) into the gingival crevice. The scores could range from 0-3 (0=Absence of inflammation; 1=Mild Inflammation-Slight change in color slight change in texture, no bleeding on probing; 2=Moderate Inflammation -glazing, redness edema and hypertrophy, bleeding on probing; 3= Severe inflammation-marked redness and hypertrophy, tendency for spontaneous bleeding)
Time Frame: Change from baseline to 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Mouthwash With Alcohol | Mouthwash Without Alcohol | Reference
Number analyzed (Participants) | 105 | 109 | 105
Units on a scale | 1.12 (0.012) | 1.11 (0.010) | 1.19 (0.014)
Statistical Analysis 1: Comparison: Mouthwash With Alcohol vs Reference; Null hypothesis that there was no difference between the two treatment groups; Test type: Superiority or Other; p < 0.0001, ANCOVA — From ANCOVA with factors for treatment group, site, smoking status, number of bleeding sites strata and the baseline GI as a covariate; Adjusted Mean Difference = -0.08, 95% CI 2-sided [-0.10 to -0.05] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Mouthwash Without Alcohol vs Reference; Null hypothesis stated that there was no difference between the two treatment groups; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Adjusted Mean Difference = -0.08, 95% CI 2-sided [-0.11 to -0.06] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Turesky Modification of Quigley & Hein Plaque Index for Overall Plaque Scores
Description: Overall plaque scores were calculated taking the average over all tooth sites for a participant. The scores could range from 0-5 (0=No plaque; 1=Slight flecks of plaque at the cervical margin of the tooth; 2= A thin continuous band of plaque (1 mm or smaller) at the cervical margin of the tooth; 3=A band of plaque wider than 1 mm but covering less than 1/3 of the area to be graded of the crown of the tooth; 4=Plaque covering at least 1/3 but less than 2/3 of the area to be graded of the crown of the tooth; 5=Plaque covering 2/3 or more of the area to be graded of the crown of the tooth)
Time Frame: Change from baseline to 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Groups:
- Reference: Brusing alone with the standard toothpaste for one timed minute twice daily for 6 weeks.
Arm/Group | Mouthwash With Alcohol | Mouthwash Without Alcohol | Reference
Number analyzed (Participants) | 105 | 109 | 105
Units on a scale | 2.50 (0.082) | 2.40 (0.084) | 3.34 (0.062)
Statistical Analysis 1: Comparison: Mouthwash With Alcohol vs Reference; Null hypothesis stated that there was no difference between the two treatment groups in Overall Plaque scores; Test type: Superiority or Other; p < 0.0001, ANCOVA — From ANCOVA with factors for treatment group, site, smoking status, number of bleeding sites strata and the baseline Plaque as a covariate; Adjusted Mean Difference = -0.80, 95% CI 2-sided [-0.98 to -0.62] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Mouthwash Without Alcohol vs Reference; Null hypothesis stated that there was no difference between the two treatment groups in Overall Plaque Scores; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Adusted Mean Difference = -0.86, 95% CI 2-sided [-1.04 to -0.68] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Turesky Modification of Quigley & Hein Plaque Index for Interproximal Plaque Scores
Description: Interproximal plaque scores were analyzed on the mesiofacial, distofacial, mesiolingual and distolingual surfaces, and calculated taking the average over all tooth sites for a participant. The scores could range from 0-5 (0=No plaque; 1=Slight flecks of plaque at the cervical margin of the tooth; 2= A thin continuous band of plaque (1 mm or smaller) at the cervical margin of the tooth; 3=A band of plaque wider than 1 mm but covering less than 1/3 of the area to be graded of the crown of the tooth; 4=Plaque covering at least 1/3 but less than 2/3 of the area to be graded of the crown of the tooth; 5=Plaque covering 2/3 or more of the area to be graded of the crown of the tooth)
Time Frame: Change from baseline to 6 weeks
Population: This analysis was conducted on ITT population, defined as those subjects who received study treatment and had at least one post-baseline efficacy measurement.
Measure: Mean (Standard Error); unit: Units on a scale
Groups:
- Mouthwash Without Alcohol: Rinse with 10ml 0.2% w/v Chlorhexidine Digluconate Mouthwash with alcohol for 1 timed minute twice daily for 6 weeks following brushing with a full brush head of standard toothpaste for 1 timed minute.
Arm/Group | Mouthwash With Alcohol | Mouthwash Without Alcohol | Reference
Number analyzed (Participants) | 105 | 109 | 105
Units on a scale | 2.77 (0.090) | 2.63 (0.091) | 3.69 (0.065)
Statistical Analysis 1: Comparison: Mouthwash With Alcohol vs Reference; Null hypotheses stated that there was no difference between the two treatments; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Adjusted Mean Difference = -0.88, 95% CI 2-sided [-1.07 to -0.69] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Mouthwash With Alcohol vs Mouthwash Without Alcohol; Null hypotheses stated that there was no difference between the two groups; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Adjusted Mean Difference = -0.97, 95% CI 2-sided [-1.16 to -0.78] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) and serious AEs were collected from the start of the washout product at visit 1, and until five days following last administration of the investigational product.
Description: The sum of number of participants affected is more than the total number affected, because multiple occurrances of an event was counted only once in a participant.
Arm/Group | Mouthwash With Alcohol | Mouthwash Without Alcohol | Reference
Serious Adverse Events (participants affected / at risk) | 0/108 | 1/109 | 0/107
Other Adverse Events (participants affected / at risk) | 67/108 | 60/109 | 47/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mouthwash With Alcohol (N=108) | Mouthwash Without Alcohol (N=109) | Reference (N=107)
Cellulitis left thigh (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mouthwash With Alcohol (N=108) | Mouthwash Without Alcohol (N=109) | Reference (N=107)
Tongue coated (Gastrointestinal disorders) | 13 (13) | 8 (8) | 2 (2)
Glossodynia (Gastrointestinal disorders) | 5 (5) | 9 (9) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 5 (6) | 6 (6) | 0 (0)
Headache (Nervous system disorders) | 19 (32) | 14 (30) | 13 (19)
Ageusia (Nervous system disorders) | 3 (3) | 6 (7) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 11 (11) | 9 (9) | 9 (9)
Dysgeusia (Nervous system disorders) | 6 (6) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 3 (5) | 2 (2) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 4 (4) | 5 (5) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 2 (2) | 5 (6) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 2 (2) | 5 (5)
Mouth injury (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) | 2 (2)
Sensitivity of teeth (Gastrointestinal disorders) | 1 (1) | 4 (4) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (3)
Oral discomfort (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Gingival injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Lip ulceration (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Oral mucosal exfoliation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Tongue disorder (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Tongue ulceration (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Traumatic ulcer (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Chapped lips (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Enlarged uvula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gingival Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gingival blister (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gingival inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tongue dry (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tongue injury (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tooth disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (4) | 2 (2)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (2) | 1 (1) | 4 (4)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (4) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (3)
Oropharyngeal pain (Reproductive system and breast disorders) | 3 (3) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (2)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Otorrhoea (Ear and labyrinth disorders) | 1 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0)
Colposcopy abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Eczema eyelids (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eye inflammation (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Limb Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.